CLINICAL TRIAL: NCT00120640
Title: Treatment of Preterm Labor With 17 Alpha-hydroxyprogesterone Caproate
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: funding
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HIC#27253
Record Dates: First submitted 2005-07-11; First posted 2005-07-18 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Premature Birth; Premature Labor
Keywords: Premature birth; Premature labor; Progesterone
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature

INTERVENTIONS:
Drug: 17 hydroxyprogesterone caproate intramuscular injections

SUMMARY:
The goal of our research will be to determine the effectiveness of 17 alpha-hydroxyprogesterone caproate (17P) in the treatment of preterm delivery. Treatment with progesterone is emerging as the standard of care for prevention of preterm delivery in asymptomatic patients at high risk for preterm birth due to a prior preterm delivery. Our goal is to evaluate whether or not progesterone is also effective in reducing preterm birth in symptomatic patients.

DETAILED DESCRIPTION:
Preterm delivery remains one of the most important issues facing perinatal medicine today. In 1999, prematurity/low birthweight accounted for 4,304 neonatal deaths, reflecting a rate of neonatal mortality due to prematurity of 23.0 per 100,000 live births. Despite the extent of the problem, the exact etiology of preterm delivery is not completely understood. It is clear that many pathways are involved in preterm delivery, and that ultimately these must converge upon one final endpoint, which is likely related to progesterone. In the animal model progesterone withdrawal is clearly directly (rodent, rabbit) or indirectly (sheep) involved in the initiation of parturition, however the exact way in which progesterone works in humans is unclear. There has been a resurgence of interest in the association between progesterone and preterm delivery. Two recent trials have looked at the utility of progesterone in the prevention of preterm delivery in high-risk patients. In a multicenter trial reported in the New England Journal of Medicine in 2003, Meis et al, recruited 463 patients with a history of spontaneous preterm delivery and randomized them in a 2:1 ratio to intramuscular 17-hydroxyprogesterone vs. placebo from 16-20 weeks until 36 weeks. Treatment with 17P significantly reduced the risk of delivery at <37 weeks, <35 weeks, and <32 weeks.

The Yale Progesterone Study is a randomized, placebo-controlled trial of the use of 17 hydroxyprogesterone for the treatment of preterm labor. The design is similar to the Meis NEJM trial, except that the patients will be symptomatic with preterm labor, rather than asymptomatic with a history of preterm delivery. In addition to the therapeutic intervention planned, the researchers intend to collect specimens to assess for markers of PTD, both before and after treatment. In this way, the researchers can analyze which pathway of PTD is involved, and finally, the effect of progesterone on these markers can be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients in preterm labor as described above.
* Patients with an accurately dated singleton gestation. Accurate dating is defined as estimated date of delivery (EDD) based on last menstrual period (LMP) dating (280 days after the first day of the LMP) confirmed by an ultrasound done before 20 weeks, which yields an EDD within 10 days of LMP dating. If the LMP is not available, the EDD must be based on 2 ultrasounds performed at least 2 weeks apart, which are concordant within 5 days of the same EDD.
* Patients with their first presentation of preterm labor will be invited to participate.
* Patients whose plan of management includes admission to the hospital and administration of antenatal steroids for fetal well being.

Exclusion Criteria:

* Rupture of membranes
* Major known fetal anomalies
* Cervical dilation > 4 centimeters
* Uterine anomalies
* Cervical cerclage
* Treatment during this pregnancy with progesterone after 14 weeks' gestation (use up to 14 weeks' gestation is permitted)
* Previous admission for preterm labor
* Contraindications to tocolysis, including fetal distress, chorioamnionitis, preeclampsia, hemodynamic instability
* Coexisting maternal disease including hypertension requiring medical therapy, cancer, seizure disorder, thromboembolic disorders, liver disease. Patients treated with oral beta adrenergics for asthma are also excluded.
* Age < 18 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-07

PRIMARY OUTCOMES:
Delivery <37 weeks' gestation
Delivery <34 weeks' gestation
Delivery <32 weeks' gestation

SECONDARY OUTCOMES:
Neonatal outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Anna K Sfakianaki, MD, Principal Investigator — Yale University; Edmund F Funai, MD, Principal Investigator — Yale University

REFERENCES:
- [Background] Meis PJ, Klebanoff M, Thom E, Dombrowski MP, Sibai B, Moawad AH, Spong CY, Hauth JC, Miodovnik M, Varner MW, Leveno KJ, Caritis SN, Iams JD, Wapner RJ, Conway D, O'Sullivan MJ, Carpenter M, Mercer B, Ramin SM, Thorp JM, Peaceman AM, Gabbe S; National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Prevention of recurrent preterm delivery by 17 alpha-hydroxyprogesterone caproate. N Engl J Med. 2003 Jun 12;348(24):2379-85. doi: 10.1056/NEJMoa035140. PMID 12802023
- [Background] da Fonseca EB, Bittar RE, Carvalho MH, Zugaib M. Prophylactic administration of progesterone by vaginal suppository to reduce the incidence of spontaneous preterm birth in women at increased risk: a randomized placebo-controlled double-blind study. Am J Obstet Gynecol. 2003 Feb;188(2):419-24. doi: 10.1067/mob.2003.41. PMID 12592250
- [Background] McLean M, Bisits A, Davies J, Woods R, Lowry P, Smith R. A placental clock controlling the length of human pregnancy. Nat Med. 1995 May;1(5):460-3. doi: 10.1038/nm0595-460. PMID 7585095